CLINICAL TRIAL: NCT05057598
Title: DianaWeb: Before and After Study Online Based Participatory Research to Test Whether Lifestyle and Diet Are Able to Reduce the Incidence of Recurrences (Local, Remote) or Secondary Cancers, Improve Prognosis and Survival of Breast Cancer
Brief Title: DianaWeb: Before and After Study Online Based Participatory Research on Breast Cancer Women
Acronym: DianaWeb
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: University Of Perugia (Other); Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other); Azienda Socio Sanitaria Territoriale di Mantova (Other); Presidio Ospedaliero Unico "Santa Maria della Misericordia", Urbino (Unknown); Ospedale Città di Castello- Perugia (Unknown); University of Urbino "Carlo Bo" (Other); Fondazione Vita e Salute (Unknown)
Responsible Party: Principal Investigator, Anna Villarini, Biologist, Nutritionist, PhD and Senior Research, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NT 24/16
Record Dates: First submitted 2021-08-28; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Diet; Physical activity; Prognosis
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Before and after study online based on community-based participatory research (CBPR): CBPR approach which has been defined as 'a process that involves community members or recipients of interventions in all phases of the research process'. Over the past two decades, there has been an increasing presence of community-based research and participatory methods in health research, and involving patients at various stages of the research process has been shown to improve the ethical nature of research and the appropriateness of methods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group on diet and lifestyles (Experimental): The arm consists to provide survivors with evidence-based recommendations and to promote improved nutrition and physical activity through videos and lectures available on the website (theoretical lectures on preventive strategies, and practical videos on cooking techniques and specific physical exercises).
  Interventions: Other: Community-based participatory research on diet and lifestyle

INTERVENTIONS:
Other: Community-based participatory research on diet and lifestyle — The intervention use a web site that contains a section to exchange information on recipes and on strategy to comply with the recommendations, and an agenda to inform on meetings, conferences, kitchen classes, walking groups, organised by the participant themselves. The investigators are developed specific recommendations for women with different characteristics. The investigators intend to improve the specificity of information with short questionnaires on portion size of relevant items using photographs or usual container in the kitchen and develop a health application for smartphone to facilitated a more efficient and timely exchange on information.
  The participants will receive a free phone number for emergencies, active 2 hours a day for 5 days a week.

SUMMARY:
DianaWeb is a community-based participatory research (CBPR) offered to Italian breast cancer patients. The aim of the study is the evaluation of effectiveness of a lifestyle and nutrition intervention to improve the prognosis. DianaWeb study utilizes an interactive website - http://www.dianaweb.org/ - to monitor patient life-style, and to obtain clinical, pathological and anthropometric data (height, body weight, waist circumference and blood pressure). Detailed instructions were provided for measuring at home. The website contains theoretical and practical advice to encourage women to follow healthy lifestyles and nutrition, and the indications emerging from research for women diagnosed with breast cancer.

DianaWeb study intends to recruit 50.000 women with breast cancer diagnosis.

DETAILED DESCRIPTION:
The investigators intend to carry out a participatory research on the influence of lifestyle after cancer diagnosis on the risk of recurrence. The investigators intend wake available to breast cancer survivors' evidence-based information on the effects of lifestyle on quality of life and prognosis and to invite and help them to adopt potentially preventive sustainable lifestyle changes. To improve the prognosis, the investigators will base the recommendations on the European Code Against Cancer 2014 (ECAC), on the World Cancer Research Fund 2018 (AICR/WCRF), Continuous Update Project (CUP) 2014 specific recommendations to breast cancer survivors, and on Mediterranean diet. As for the prevention of side effect of treatments there is no definitive evidence, but the daily exercise seems for reducing menopausal symptoms and osteoporosis, while regular consumption of food with diuretic effect for arthralgia due to aromatase inhibitors. The investigators are aware that the path for creating data to implementing evidence in routine practice is long and arduous. The investigators are confident, however, that engaging participants in the research process will enable many of participants to implement evidence-based practices in everyday life. The investigators, together with computer programmers, have developed an interactive website to build a large cohort of breast cancer survivors and to follow up participants about the impact of lifestyles and nutrition on recurrences, incidence of second breast cancer, metastasis, other cancers and other chronic diseases. The investigators will also monitor the prevalence of side effects of treatments (the investigators will focus on menopausal symptoms, arthralgia, osteoporosis and bone fractures). Observational epidemiological studies have consistently shown that sedentary lifestyle, overweight, metabolic syndrome, chronic inflammatory status, high glycemia and insulinemia, and a few specific dietary factors (low fibre and high saturated fat) are associated with poor breast cancer specific survival. There is ample room for reducing recurrences and cancer progression through lifestyles and nutrition. All these factors are clearly modifiable, but there is uncertainty, however, over whether voluntarily changing these factors after breast cancer diagnosis improve prognosis. In a 5 years' time the study after recruitment, the investigators are expected to confirm the prognostic role of this factors.

In Italy every year over 50.000 women develop breast cancer. The country is fairly well equipped with excellent breast cancer units and in the second decade of the twenty-first century 5-year breast cancer net survival reached 88%, a performance similar to the best European countries. Over 750.000 Italian women live with a previous diagnosis of breast cancer. Many of them with some form of cancer treatment and suffer from feeling left alone, fear of cancer recurrence and not receiving enough information and guidance after treatment: on prognosis, side effects of treatment, lifestyle strategies to help preventing side effects of treatments, recurrences and new primaries. Many survivors integrate adjuvant treatment with complementary treatments without scientific proof of efficacy, even with folk treatments that might increase the risk of recurrences.

Young women undergoing adjuvant breast cancer therapy experience a heavy impairment in important quality of life domains (anxiety, depression, loss or sexual desire, weight gain). The great majority of women under hormonal treatment experience an increase in the prevalence of menopausal symptoms and have sexual dysfunction that is distressing and difficult to resolve. In postmenopausal survivors with aromatase inhibitor-induced arthralgia the intensity of pain is associated with fear of recurrence.

Investigating whether lifestyle factors affect breast cancer patients' survival is a relatively new area of research, but there is growing evidence that the effect of modifiable anthropometric and metabolic factors may be of the same order of magnitude than the effect of the usual clinic-pathological risk factors.

Epidemiological evidence, even if based only on observational studies, suggest that lifestyle modification, including physical exercise and dietary habits, might have a strong impact on breast cancer patients overall and specific survival.

CUP have shown that:

1. overweight and obesity are associated with 10-20% increased risk of recurrences;
2. physical activity after diagnosis is associated with 30-40% reduction of recurrences and mortality;
3. soy food consumption is associated with lower risk
4. saturated fat consumption is associated with higher risk
5. higher consumption of foods containing fibre after diagnosis of primary breast cancer reduces risk of all-cause mortality Epidemiological studies have shown that modifiable lifestyle factors and biomarkers affecting the occurrence of breast cancer also affect breast cancer prognosis: obesity, metabolic syndrome, sedentary lifestyle, high fat intake, alcohol consumption, high fasting glucose plasma levels (independently of the presence of metabolic syndrome), clinical chronic inflammation, high plasma insulin and sex hormone levels, low sex hormone-binding protein.

Obesity is associated with a higher incidence of locally advanced disease, and worse prognosis after diagnosis, both before and after menopause.

The obesity is also related to poor quality of life and increased risk of developing comorbid conditions. Weight gain during and after cancer treatment also increases the risk of recurrence. Both chemotherapy and, to a lesser extent, tamoxifen and nonsteroidal aromatase inhibitors have been associated with weight gain. Among the potential mechanisms behind the association between weight gain, obesity, and breast cancer recurrence and mortality there is an increased conversion of androgens to oestrogens in peripheral adipose tissue and increased circulating levels of insulin, insulin-like growth factors (IGFs), and leptins, that promote tumour cell proliferation. Current breast cancer treatments can have a negative impact on cardiovascular health (left ventricular dysfunction, accelerated cardiovascular disease-CVD), and for women with pre-existing CVD, this might influence cancer treatment decisions by both the patient and the provider. Improvements in early detection and treatment of breast cancer have led to an increasing number of breast cancer survivors who are at risk of long-term cardiac complications from cancer treatments. Ideal breast cancer outcomes are reliant on coexisting cardiovascular health along the entire journey of breast cancer treatment. During breast cancer treatment, surveillance, prevention, and secondary management of cardiotoxicity are crucial; thereafter, long-term post-treatment monitoring for late cardiotoxicity and even non-treatment-related development of CVD is essential. Breast cancer and CVD share a number of common risk factors. Cardiovascular clinical care and research have focused on risk factors for >60 years, because it is believed that 80% of CVD can be prevented through risk factor modifications such as promoting a healthy diet, physical activity, and a healthy weight; abstinence from tobacco; blood pressure control; diabetes mellitus management; and a good lipid profile. In women with breast cancer, treatment and the disease itself contribute to weight gain and to decreases in physical activity. Furthermore, it has been reported that cardiopulmonary function in patients with breast cancer improves with exercise, and regular exercise results in an improvement in quality of life. Although the usefulness of exercise to prevent CVD in patients with breast cancer has not been evaluated in randomized trials, it is reasonable to follow the recommendations for physical activity, that is, moderate-intensity aerobic physical activity of ≥30 minutes 5 days each week.

High fasting glycaemia, even within the normal range, is associated with higher incidence of recurrences. Also, the metabolic syndrome is associated with increased risk of breast cancer recurrences in patients diagnosed both before and after menopause and risk of developing distant metastasis than patients without any metabolic syndrome trait. Metabolic syndrome, also called insulin-resistance syndrome, is usually associated with high insulin and testosterone levels, and with clinical chronic inflammation. Independently of the presence of metabolic syndrome several studies have shown that breast cancer patients with high testosterone levels have worst prognosis. Insulin stimulates the synthesis of testosterone in the ovary, and high plasma insulin levels are associated with increased risk of recurrences. Insulin also increases the bioavailability of IGF-I (through the promotion of its liver synthesis and the inhibition of the synthesis of its binding proteins IGFBP-I) associated with prognosis in women with breast cancer. Also, high plasma levels of C-Reactive Protein (CRP), even within the normal range, are associated with increased risk of recurrence and shorter survival in patients with advanced breast cancer. It seems reasonable to hypothesize that a comprehensive lifestyle modification, based on AICR/WCRF and ECAC recommendations, consistent with traditional Mediterranean diet, may reduce the risk of recurrences and improve prognosis. Studies have shown that dietary intervention recommending a modified Mediterranean diet can reduce biological markers of breast cancer risk and recurrences: glycemia, insulinemia, IGF-I bioavailability and chronic inflammatory status. The Western dietary pattern, high in refined grains, sugars, simple carbohydrates, red meat, and high-fat dairy products, increases the levels of pro-inflammatory markers such as CRP and interleukin-6 (IL-6). In contrast, a traditional Mediterranean diet with consumption of whole grains cereals, pulses, vegetables, fruits, fish, nuts and extravirgin olive oil is associated with lower levels of pro-inflammatory biomarkers, including endothelial adhesion molecules, CRP, and tumor necrosis-α (TNF-α). Physical exercise also seems to reduce chronic inflammation. Furthermore, several studies have suggested a decrease of breast cancer recurrence and death in patients who exercise at least 30 min /day.

These information's are not currently available to patients and are not yet included in oncology protocols. With a few exceptions, physicians too are not aware of these scientific results and are not yet culturally prepared for life-style prescriptions. DianaWeb does not interfere with prescribed oncological treatments, on the contrary it recommends participants to follow the oncologist's prescriptions, but the study wants avoid the access to non-scientifically correct information that could worsen the prognosis or change the quality of life or health.

There is increasing interest, in the research community, in a community-based participatory research. Its relevance often is relegated to the "right end" of the research continuum, but may contribute also to asking the right questions, in particular the more relevant questions for the patients, to improve compliance, and to ensure that basic science research findings affect cancer outcomes in materially important ways especially for large communities that communicate through modern media as websites.

ELIGIBILITY:
Inclusion Criteria:

* Women with breast cancer diagnosis
* Women with breast cancer relapses
* Women with breast cancer metastases
* Women with breast cancer diagnosis even if many years have elapsed since the first diagnosis
* Women with breast cancer diagnosis and other tumors diagnosis
* Women with breast cancer diagnosis and other pathologists that impair cognitive abilities

Exclusion Criteria:

* Women with breast cancer diagnosis and clinical diagnosis of Alzheimer's Disease
* Women with breast cancer diagnosis and clinical diagnosis of dementia
* Women with breast cancer diagnosis unable to use personal computer and smart phone

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with breast cancer diagnosis
Enrollment: 50000 (Estimated)
Dates: Start 2016-06-21 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Increase rate of survival | Baseline, 10 years
  Evaluate the change in rate of survival in relation to adherence to correct lifestyles and health nutrition (ECAC, AICR/WCRF recommendations and Mediterranean diet) through the information provided by the family members, the physician and the cancer registry.
Decrease incidence of relapses | Baseline, 10 years
  Evaluate the change about incidence of relapses in relation to adherence to correct lifestyles and health nutrition (ECAC, AICR/WCRF recommendations and Mediterranean diet) through the information provided by the patient and the physician.
Decrease incidence of metastasis | Baseline, 10 years
  Evaluate the change about incidence of metastasis in relation to adherence to correct lifestyles and health nutrition (ECAC, AICR/WCRF recommendations and Mediterranean diet) through the information provided by the patient and the physician.
Decrease incidence of Metabolic Syndrome parameters | baseline, 1 year, 5 years, 10 years
  Evaluate the change about incidence of Metabolic Syndrome parameters in relation to adherence to correct lifestyles and health nutrition (ECAC, AICR/WCRF recommendations and Mediterranean diet).
Decrease blood level on C-reactive protein (chronic inflammation marker) | baseline, 1 year, 5 years, 10 years
  Evaluate the change of the blood level on C-reactive protein, in relation to adherence to correct lifestyles and health nutrition (ECAC, AICR/WCRF recommendations and Mediterranean diet).
Decrease the insulin resistance index (HOMA index) | baseline, 1 year, 5 years, 10 years
  Evaluate the change in the insulin resistance index, in relation to adherence to correct lifestyles and health nutrition (ECAC, AICR/WCRF recommendations and Mediterranean diet).

SECONDARY OUTCOMES:
Increase in the score of adherence to the Mediterranean diet score (MDS) | baseline, 1 year, 3 years, 5 years, 10 years
  Evaluate the change about Mediterranean diet through the use of the MDS: Low adhesion 0-3; Average adhesion 4-5; High adhesion 6-9.
Increase in the score of adherence to the Italian Mediterranean index (IMI) | baseline, 1 year, 3 years, 5 years, 10 years
  Evaluate the change about Italian Mediterranean index through the use of the IMI: Low adhesion 0-1; Fair adhesion 2-3; Good adhesion 4-5; High adhesion 6-11.
Increase in the score of adherence to the Mediterranean Adequancy index (MAI) | baseline, 1 year, 3 years, 5 years, 10 years
  Evaluate the change about Italian Mediterranean index through the use of the MAI: the higher the percentage number the greater the adhesion to the index.
Increase in the score of adherence to the AICR/WCRF recommendations to the 2018 WCRF/AICR News Score | baseline, 1 year, 3 years, 5 years, 10 years
  The 2018 WCRF/AICR Cancer Prevention Recommendations, goals, and statements of advice were examined to define components of the New Score. Eight of the ten 2018 WCRF/AICR Recommendations concerning weight, physical activity, diet, and breastfeeding (optional), were selected for inclusion. Each component is worth one point: 1, 0.5, and 0 points for fully, partially, and not meeting each recommendation, respectively (Score: 0 to 7-8 points). Two recommendations on dietary supplement use and for cancer survivors are not included due to operational redundancy.
Increase in the score to the "European Organisation for Research and Treatment of Cancer, Quality of Life questionnaire-core 30 (Version 3.0)" after breast cancer diagnosis | baseline, 1 year, 3 years, 5 years, 10 years
  Test the hypothesis that participation in a community of women with breast cancer improve quality of life through QLQ-C30: is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. The single item measures range in score from 1 to 4 (28 items) and from 1-7 (2 items).
  A high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL (max 14), but a high score for a symptom scale / item represents a high level of symptomatology / problems (max 112).
Increase in the score to the "European Organisation for Research and Treatment of Cancer, Quality of Life questionnaire-breast cancer 45 (QLQ-BR45)" during therapy | baseline, 1 year, 3 years, 5 years, 10 years
  Test the hypothesis that participation in a community of women with breast cancer improve quality of life through QLQ-BR45. The EORTC has already validated the QLQ-BR23, a questionnaires developed to assess quality of life (QoL) in patients with breast cancer (BC). The new module contains a total of 45 items, 23 items from the BR 23 and 22 new items: 23 questions assessing disease symptoms, side effects of treatment (surgery, chemotherapy, radiotherapy and hormonal treatment), body image, sexual functioning and future perspective and 2 multi-item scales: target symptom scale (20 items divided in 3 subscales: endocrine therapy scale, endocrine sexual scale and skin/mucosa scale) and satisfaction scale (2 items). The scoring approach for the QLQ-BR45 is identical in principle to that for the function and symptom scales / single items of the QLQ-C30.

CONTACTS AND LOCATIONS:
Overall Officials: ANNA VILLARINI, PhD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano
Locations (1):
- Fondazione Irccs Istituto Nazionale Dei Tumori, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, dataset, statistical analysis plan, informed consent form and clinical study report were discussed through meetings held with all the collaborating centers. The individual participant data (IPD) were delivered to the coordinators of the individual centers in coded anonymous.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be become available from baseline up to 10 years after study the end of recruitment for all coordinators of collaborating centers
Access Criteria: The data are available on the National Cancer Institute of MILANO (Foundation-Institute of Hospitalization and Scientific Care), network managed

REFERENCES:
- [Result] Natalucci V, Marini CF, Flori M, Pietropaolo F, Lucertini F, Annibalini G, Vallorani L, Sisti D, Saltarelli R, Villarini A, Monaldi S, Barocci S, Catalano V, Rocchi MBL, Benelli P, Stocchi V, Barbieri E, Emili R. Effects of a Home-Based Lifestyle Intervention Program on Cardiometabolic Health in Breast Cancer Survivors during the COVID-19 Lockdown. J Clin Med. 2021 Jun 17;10(12):2678. doi: 10.3390/jcm10122678. PMID 34204528
- [Result] Natalucci V, Villarini M, Emili R, Acito M, Vallorani L, Barbieri E, Villarini A. Special Attention to Physical Activity in Breast Cancer Patients during the First Wave of COVID-19 Pandemic in Italy: The DianaWeb Cohort. J Pers Med. 2021 May 6;11(5):381. doi: 10.3390/jpm11050381. PMID 34066580
- [Result] Gianfredi V, Nucci D, Balzarini M, Acito M, Moretti M, Villarini A, Villarini M. E-Coaching: the DianaWeb study to prevent breast cancer recurrences. Clin Ter. 2020 Jan-Feb;170(1):e59-e65. doi: 10.7417/CT.2020.2190. PMID 31850486
- [Result] Villarini M, Acito M, Gianfredi V, Berrino F, Gargano G, Somaini M, Nucci D, Moretti M, Villarini A. Validation of Self-Reported Anthropometric Measures and Body Mass Index in a Subcohort of the DianaWeb Population Study. Clin Breast Cancer. 2019 Aug;19(4):e511-e518. doi: 10.1016/j.clbc.2019.04.008. Epub 2019 Apr 18. PMID 31182401
- [Result] Villarini M, Lanari C, Nucci D, Gianfredi V, Marzulli T, Berrino F, Borgo A, Bruno E, Gargano G, Moretti M, Villarini A. Community-based participatory research to improve life quality and clinical outcomes of patients with breast cancer (DianaWeb in Umbria pilot study). BMJ Open. 2016 Jun 1;6(6):e009707. doi: 10.1136/bmjopen-2015-009707. PMID 27251681

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT05057598/Prot_SAP_000.pdf